CLINICAL TRIAL: NCT00622752
Title: A Double-Blind, Randomized, Placebo- and NRT -Controlled Phase II Study to Assess the Effects of EVT 302 Alone and in Combination With NRT on Craving and Withdrawal in Healthy Male Smokers Deprived of Cigarettes
Brief Title: Effects of EVT 302 With or Without NRT on Craving and Withdrawal in Healthy Male Smokers Deprived of Cigarettes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evotec Neurosciences GmbH (Industry)
Responsible Party: Doris Greiling, Clinical Development Programme Manager, Evotec Neurosciences GmbH
Organization: Evotec International GmbH (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EVT 302/3011; EUDRACT No.: 2007-006236-63
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Craving; Smokers
MeSH Terms: conditions — Smoking Cessation | interventions — sembragiline; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): EVT 302, 10 mg
  Interventions: Drug: EVT 302, 10 mg
- 2 (Experimental): EVT 302, 10 mg + NRT patch, 21 mg
  Interventions: Drug: EVT 302, 10 mg; Drug: Nicotine replacement therapy (NRT)
- 3 (Experimental): NRT patch, 21 mg
  Interventions: Drug: Nicotine replacement therapy (NRT)
- 4 (Placebo Comparator): Placebo to match EVT 302 and placebo patch to match NRT patch
  Interventions: Drug: placebo; Device: NRT placebo

INTERVENTIONS:
Drug: EVT 302, 10 mg — 2 X EVT 302, 5 mg tablets
  Arms: 1; 2
Drug: placebo — 2 X placebo tablets to match EVT 302 5 mg
  Arms: 4
Drug: Nicotine replacement therapy (NRT) — NRT patch containing 21 mg of nicotine
  Arms: 2; 3
Device: NRT placebo — Medically inert plaster cut to match the NRT plaster
  Arms: 4

SUMMARY:
This randomised, placebo-controlled study is designed to explore the effects of EVT 302 both with and without concomitant nicotine replacement therapy (NRT) on craving and withdrawal in smokers after short term deprivation of cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 18 and 55 years of age, inclusive
* BMI between 18 and 30, minimum weight of 50 kg
* Negative urine drug & alcohol screen
* Able to comply with tyramine-restricted diet
* Smoking of ≥17 and ≤34 cigarettes per day for the past year and have not tried to quit smoking in the 3 months prior to screening
* Subjects are willing and able to quit for about 12 hours in each of three subsequent study periods
* Previous experience of craving following smoking cessation
* Breath CO between 15 ppm and 20 ppm and cotinine in saliva and plasma at least 250 ng/mL at screening
* Liver function test results not above 1.5 times the upper normal limit (UNL) at screening visit and at re-assessment during the study.

Exclusion Criteria:

* Participation in another clinical study within 60 days of screening
* Evidence of active significant psychiatric or neurological disease or dependency other than cigarettes
* Are known to have or are a carrier of the hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, has a positive result to the human immunodeficiency virus-1 and/or 2 (HIV-1 and/or HIV-2) antibodies
* Known hypersensitivity to MAO inhibitors or any substance that is contained in the study formulations
* Known allergy to plasters or NRT patches
* Previous participation in another study with EVT 302
* Currently receiving treatment for smoking cessation
* Current use of tobacco products other than cigarettes
* Require treatment with any medication
* Subject with a clinically relevant abnormal 12-lead ECG recording or QTcB/F >430 ms
* Use of a prescription medicine within 14 days or 5 half-lives, whichever is the longer, of the start of dosing, or use of an over-the-counter medication during the 7 days before the study, including herbal remedies, but excluding paracetamol and vitamin supplements (provided intake does not exceed the daily recommended allowance)
* Subjects must not be planning to father a child or donate sperm, during the study and 3 months after the end of the study. Acceptable methods of contraception comprise barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least 2 month)
* Daily consumption of more than 5 cups of tea or coffee, or more than 1.0 litre of xanthine-containing drinks
* Recent myocardial infarction, unstable or worsening angina pectoris, prince metal angina, severe arrhythmias, recent stroke.
* Creatinine clearance (CLR) calculated according to the formula by Modification of Diet in Renal Disease (MDRD) of <80 mL/min

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Reduction in Craving and withdrawal | Within 12 hours of the last cigarette

SECONDARY OUTCOMES:
CogState Cognitive test Battery | 12 hours post last cigarette
Breath carbon monoxide levels | 12 hours post last cigarette
Salivary cotinine levels | 12 hours post last cigarette
Clinical safety lab tests | Up to 7 days post dose
Assessment of adverse events | Up to 7 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Alla Radicke, MD, Principal Investigator — Parexel International GmbH, Clinical Pharmacology Research Unit
Locations (1):
- PAREXEL International GmbH, Clinical Pharmacology Research Unit, Berlin, Germany